CLINICAL TRIAL: NCT06655636
Title: Assisting Stroke Survivors With Engineering Technology (ASSET): Design Project D3: Exoskeletal Networks for Forearm Supination
Brief Title: Safety and Feasibility of an ExoNET for Supination Assistance for Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Co-Director, Robotics Laboratory, Arms and Hands Lab, Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00218538
Record Dates: First submitted 2024-03-25; First posted 2024-10-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Cerebral Vascular Accident
Keywords: Upper Extremity; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Assistance, Sham, Anti-Assistance (Experimental): Group 1 receives all three interventions in the order of assistance, then sham (slack springs), then anti-assistance. Each intervention corresponds to different settings on the device.
  Interventions: Device: Device tuned to Assistance; Device: Device tuned to Sham (Slack Springs); Device: Device tuned to Anti-Assistance
- Group 2 - Sham, Assistance, Anti-Assistance (Experimental): Group 2 receives all three interventions in the order of sham (slack springs), then assistance, then anti-assistance. Each intervention corresponds to different settings on the device.
  Interventions: Device: Device tuned to Assistance; Device: Device tuned to Sham (Slack Springs); Device: Device tuned to Anti-Assistance

INTERVENTIONS:
Device: Device tuned to Assistance — The device spring components will be tuned to produce an assistive supination torque on the forearm.
Device: Device tuned to Sham (Slack Springs) — The device spring components will be tuned to slack springs to serve as a placebo. The user will think they are receiving forces but in reality the device will not be providing any forces.
Device: Device tuned to Anti-Assistance — The device spring components will be tuned to produce a resistive supination torque on the forearm.

SUMMARY:
The purpose of this study is to evaluate the safety, feasibility, and efficacy of an exoskeletal network of passive, multi-joint springs for forearm supination. Also known as the forearm ExoNET, the device is a passive, robotic device that will properly assist forearm supination in the post-stroke adult population.

DETAILED DESCRIPTION:
The ExoNET, a passive robotic solution that provides a soft, biomimetic, and elastic alternative to robotics that embodies intelligence within the mechanical design. Several groups have been exploring performance enhancement using springs with custom-tuned parameters via optimization. Here, it is possible to have a simple reconfigurable system that can not only assist performance, but can also make training easier, faster, and more complete. This contribution has the potential to be clinically significant for rehabilitating neurologically impaired individuals because this proposal will investigate how motor learning can be facilitated through novel assistive technology.

The primary objective of this study is to evaluate the safety, feasibility, and efficacy of using the forearm ExoNET. Specifically, investigators would like to see if the forearm ExoNET tuned to assistance will lead to a reduction in forearm muscle activity and an increase in active supination range of motion. To accomplish this, we plan to have participants perform upper extremity activities of daily living requiring active forearm supination wearing the ExoNET. To achieve these goals, we will use a wearable surface electromyography (EMG) and inertial measurement unit (IMU) using Delsys wearable sensors on the forearm muscles.

Investigators hypothesize that individuals with post-stroke arm movement deficits will experience gains in Action Research Arm Test (ARAT) measures that are significantly above their baseline levels while using the forearm ExoNET tuned to supination assistive support. Secondarily, investigators hypothesize that a forearm ExoNET tuned to supination assistive support will lead to a significant reduction in arm muscle activity and no significant difference in range of motion across a series of upper-extremity tasks in adults without a history of stroke. Lastly, it is hypothesized that usage of a forearm ExoNET tuned to supination anti-assistance can be safe, feasible and tolerated by patients in a given treatment session.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 40-70 (to reduce confounding effects of aging on muscle, movement accuracy and proprioception)
2. Have sustained a single, unilateral stroke at least 8 months prior to enrollment
3. Severe to moderate upper extremity impairment (ARAT score 0-30)
4. Ability to move their elbow and wrist when supported against gravity
5. Cortical stroke with hemiparesis, tactile sensation
6. Available medical records about lesion locations indicating the stroke was caused by a middle cerebral artery ischemic infarct

Exclusion Criteria:

1. Bilateral paresis
2. Diffuse/multiple lesion sites or multiple stroke events
3. Hemispatial neglect or visual field cut that prevent visual feedback
4. Shoulder pain and/or articular rigidity on the upper limb joint
5. Severe sensory deficits indicated by the Two-Point Discrimination Test
6. Botox injection to the affected upper extremity within the previous 4 months
7. Aphasia, cognitive impairment, or affective dysfunction that would influence the ability to consent, perform the experiment, or follow commands
8. Concurrent participation in upper extremity rehabilitation either as part of a research intervention protocol or a prescribed therapy
9. Other neurological issues
10. Meet any of the contraindications to Delsys Trigno Sensors:

    * Implanted with electronic devices of any kind, including cardiac pace-makers or similar assistive devices, electronic induction pumps, and implanted stimulators
    * Irritated skin or open wounds
    * Silver allergy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Tested at week 1 (baseline evaluations), week 2 (post evaluation), week 3 (post evaluation)
  Observational measure used to assess change in upper extremity performance in individuals with a damaged nervous system

SECONDARY OUTCOMES:
Upper extremity portion of the Fugl-Meyer (FMUE) | Tested at week 1 (baseline evaluations), week 2 (post evaluation), week 3 (post evaluation)
  Observational measure used to measure change in upper extremity impairment in individuals with a damaged nervous system
Box and Blocks | Tested at week 1 (baseline evaluations), week 2 (post evaluation), week 3 (post evaluation)
  Measures change in unilateral gross motor dexterity

OTHER OUTCOMES:
Electromyography using Delsys | Treatment phases (week 1, week 2 and week 3)
  Delsys sensors will be used to measure change in biceps activity
Joint Kinematics using Microsoft Kinect | Treatment phases (week 1, week 2 and week 3)
  Markerless joint tracking system will be used to collect changes in the joint kinematics to identify changes in limb movement compensatory strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lannin NA, Cusick A, Hills C, Kinnear B, Vogel K, Matthews K, Bowring G. Upper limb motor training using a Saebo orthosis is feasible for increasing task-specific practice in hospital after stroke. Aust Occup Ther J. 2016 Dec;63(6):364-372. doi: 10.1111/1440-1630.12330. Epub 2016 Sep 19. PMID 27646624
- [Background] Gijbels D, Lamers I, Kerkhofs L, Alders G, Knippenberg E, Feys P. The Armeo Spring as training tool to improve upper limb functionality in multiple sclerosis: a pilot study. J Neuroeng Rehabil. 2011 Jan 24;8:5. doi: 10.1186/1743-0003-8-5. PMID 21261965
- [Background] J. S. Sulzer, M. A. Peshkin and J. L. Patton, "MARIONET: An exotendon-driven rotary series elastic actuator for exerting joint torque," 9th International Conference on Rehabilitation Robotics, 2005. ICORR 2005., Chicago, IL, USA, 2005, pp. 103-108, doi: 10.1109/ICORR.2005.1501062.
- [Background] Ryali, P., Carella, T., McDermed, D., Perizes, V., Huang, F., & Patton, J. (2020). A Theoretical Framework for a Network of Elastic Elements Generating Arbitrary Torque Fields. In 2020 8th IEEE RAS/EMBS International Conference for Biomedical Robotics and Biomechatronics (BioRob) (pp. 286-291). IEEE.